CLINICAL TRIAL: NCT06923254
Title: 7.0T Magnetic Resonance Imaging Study for Hepatic Encephalopathy
Status: Not yet recruiting | Type: Observational
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Xin Lou, Deputy Director of Department of Radiology, Chinese PLA General Hospital
Other Study IDs: Hepatic encephalopathy-301
Record Dates: First submitted 2025-04-04; First posted 2025-04-11 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: Hepatic Encephalopathy (HE); MRI; fMRI Research
Keywords: Hepatic Encephalopathy; fMRI
MeSH Terms: conditions — Hepatic Encephalopathy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- 7.0T Research: With the advantages of 7.0TMRI, we detect the imaging characteristics of patients with hepatic encephalopathy (HE).
  Interventions: Other: 7.0T MRI-Scan

INTERVENTIONS:
Other: 7.0T MRI-Scan — 7.0T MRI-Scan

SUMMARY:
This clinical trial study aims to detect the imaging characteristics of patients with hepatic encephalopathy (HE) using 7-Tesla (7T) magnetic resonance imaging (MRI).

DETAILED DESCRIPTION:
In this study, we analyzed the imaging characteristics of HE. First, with the advantages of 7TMRI, we analyzed the differences in imaging characteristics between HE patients and the healthy, including brain functional imaging and structural imaging. Second, we analyzed the differences in imaging characteristics between different subgroups of HE patients. Finally, we analyzed the correlation between the prognostic results of HE patients after follow-up and the imaging characteristics.

ELIGIBILITY:
Inclusion Criteria:

* Patients with clinical suspected or diagnosed hepatic encephalopathy according to relevant guidelines.The patient's education level is above primary school level.
* Regular follow-up.

Exclusion Criteria:

* Contraindications to MRI.
* Patients with cerebrovascular disease, brain tumors, epilepsy, other neurodegenerative disease.

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with hepatic encephalopathy
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-04-03 (Estimated); Primary Completion 2029-12-24 (Estimated); Study Completion 2030-12-24 (Estimated)

PRIMARY OUTCOMES:
Functional connectivity and structural alterations between individuals with different subtypes of HE and healthy subjects. | 5 years
  Functional connectivity calculation is mainly based on the BOLD sequence, which is used to describe the degree of connectivity between different brain regions and reflect the functional activity of the brain. Gray matter (GM) morphological destruction, cortical thickness, and subcortical nuclear volume in patients with hepatic encephalopathy were analyzed based on structural magnetic resonance imaging（sMRI）.

SECONDARY OUTCOMES:
Correlation between spectral features of clinical variables and spectral features of imaging. | 5 years
  The clinical variable spectrum characteristics were constructed using the patients' medical records and test data. The distribution characteristics of clinical psychological characteristics and imaging spectrum characteristics were compared using a multidimensional matrix, and gene-imaging association analysis was used to evaluate imaging changes.

CONTACTS AND LOCATIONS:
Overall Officials: Xin Lou, Study Chair — Chinese PLA General Hospital
Locations (1):
- Chinese PLA General Hospital, Beijing, Beijing Municipality, China